CLINICAL TRIAL: NCT02427945
Title: Leveraging an Existing Large-scale Safe Water Program to Deliver Nutrition Messages at a Low Marginal Cost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcos Vera Hernandez (Other)
Collaborators: Evidence Action (Unknown); MaiMwana (Unknown)
Responsible Party: Sponsor-Investigator, Marcos Vera Hernandez, Research Fellow, Institute for Fiscal Studies
Organization: Institute for Fiscal Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1827/006
Record Dates: First submitted 2015-04-14; First posted 2015-04-28 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Child Malnutrition
Keywords: Information provision
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Child Nutritional Physiological Phenomena

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Provision of information on safe water
  Interventions: Behavioral: Provision of information on safe water
- Treatment traditional (Experimental): Provision of information on safe water and child nutrition. The information will be targeted to the mother of the child aged between 6 and 24 months old.
  Interventions: Behavioral: Provision of information on safe water and child nutrition
- Treatment couple (Experimental): Provision of information on safe water and child nutrition. The information will be targeted to the mother of the child aged between 6 and 24 months old, and her husband.
  Interventions: Behavioral: Provision of information on safe water and child nutrition

INTERVENTIONS:
Behavioral: Provision of information on safe water — A promoter from Evidence Action will visit the household and provide information on safe water.
  Arms: Control
Behavioral: Provision of information on safe water and child nutrition — A promoter from Evidence Action will visit the household and provide information on safe water, as well as child nutrition (including hygiene on food preparation and storage). Households will be given a poster to hang in their dwellings with basic nutrition information. The poster might be smaller and in black and white, or larger and in color.
  Arms: Treatment couple; Treatment traditional

SUMMARY:
The investigators are seeking to overcome the dual challenges of under-nutrition and diarrhea using an existing safe water supply platform to deliver nutrition information to targeted groups in Western Kenya. Using a randomized evaluation, investigators will determine the impact on nutrition status and practices of delivering nutrition information. The evaluation results will enable Evidence Action to make strategic decisions regarding the potential scale-up of the combined program across Kenya.

DETAILED DESCRIPTION:
Evidence Action's Dispensers for Safe Water program currently provides access to safe water for two million people. The program would be able to leverage the existence of this service delivery platform to provide promoters with training on proper nutrition and methods for delivering these messages to target groups.

The intervention is a home visiting program that will provide nutrition advice on complementary feeding to households with children aged 6-24 months. Two types of home visits will be evaluated, a 'traditional visit mode' in which the child's mother receives the visit; and a 'couples visit mode' in which the promoter attempts to involve both the father and mother.

Households in the control group will also receive home visits by promoters but the content of the visit will be restricted to safe water. The same information on safe water will also be provided to households in the treatment group. Hence, the evaluation will measure the additional effect of providing nutrition information on top of information on safe water.

Promoters will provide advice on nutrition and food hygiene to target households, according to criteria established by Evidence Action. Following the Guiding Principles for Complementary Feeding of the Breastfed Child (PAHO/WHO 2003), the intervention will include information on the maintenance of breastfeeding, safe/hygienic preparation and storage of complementary foods, amount of complementary food needed, food consistency, meal frequency and energy density, nutrient content of complementary foods, and feeding after illness. The home visits will be modelled on the MaiMwana Infant Feeding intervention (http://www.maimwana.malawi.net/MaiMwana/Home.html) that has been taking place in Mchinji (Malawi) since 2005.

Households within the treatment group will be provided by a poster to hang in their dwellings with some basic information on nutrition. A random subset of households will be given a small poster in black and white, and the other subset of households will be give a larger color poster.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included if they are between 0 and 18 months at baseline and live within the catchment area of a water point in which Evidence Action installs a chlorine dispenser

Exclusion Criteria:

* None

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1671 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Height-for-age z-score | Up to 18 months

SECONDARY OUTCOMES:
Knowledge of child nutrition issues measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Child nutritional intake measured using a 7 day Food Frequency Questionnaire | Up to 18 months
  Measured using a 7 day Food Frequency Questionnaire
Child's age when breastfeeding stops measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
A composite index of other anthropometric indicators (includes child's weight for age z-score, child's mid-upper arm circumference, and child's head circumference) | Up to 18 months
  The composite index will include child's weight for age z-score, child's mid-upper arm circumference, and child's head circumference.
Probability that the child suffers from bipedal oedema | Up to 18 months

OTHER OUTCOMES:
Household food consumption measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Household consumption measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Total Chlorine Residual score | Up to 18 months
Labor supply measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Time cooking on the day prior to the interview measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Women's empowerment measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire
Probability of having a chat with a friend or acquaintance about food or nutrition measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire. Having a chat in the last 3 days prior to the survey interview.
Probability of child suffering from diarrhea measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire. Suffering from diarrhea in the last 7 days prior to the survey. Diarrhea is defined as having 3 loose stools in any one day and/or having blood in the stools at least once.
Hygiene practices measured using a structured questionnaire | Up to 18 months
  Measured using a structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Vera-Hernandez, PhD, Principal Investigator — Research Fellow
Locations (1):
- Evidence Action, Busia, Busia County, Kenya